CLINICAL TRIAL: NCT07381738
Title: A Single-arm, Two-center, Prospective Clinical Study of Unrelated Cord Blood Transplantation for EBV-associated Lymphoproliferative Disorders
Brief Title: Unrelated Cord Blood Transplantation for EBV-associated Lymphoproliferative Disorders
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Fudan University (Other)
Collaborators: Huashan Hospital (Other)
Responsible Party: Principal Investigator, Zhijun Bao, Director, Fudan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2025K399
Record Dates: First submitted 2026-01-20; First posted 2026-02-02 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Epstein-Barr Virus-associated Lymphoproliferative Diseases; Chronic Active Epstein-Barr Virus Infection; EBV Associated Lymphoma; Umbilical Cord Blood Transplant
Keywords: Epstein-Barr virus-associated lymphoproliferative diseases; Chronic Active Epstein-Barr Virus Infection; EBV Associated Lymphoma; Umbilical Cord Blood Transplant

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment arm (Experimental): All participants will be enrolled in the treatment group and will receive a standard-dose unrelated cord blood transplantation. The efficacy and safety of unrelated cord blood transplantation for the treatment of Epstein-Barr virus-associated lymphoproliferative diseases will be evaluated.
  Interventions: Procedure: Umbilical cord blood transplantation as treatment of Epstein-Barr virus-associated lymphoproliferative diseases

INTERVENTIONS:
Procedure: Umbilical cord blood transplantation as treatment of Epstein-Barr virus-associated lymphoproliferative diseases — All participants will be enrolled in the treatment group and will receive a standard-dose unrelated cord blood transplantation. The efficacy and safety of unrelated cord blood transplantation for the treatment of Epstein-Barr virus-associated lymphoproliferative diseases will be evaluated.

SUMMARY:
This clinical trial is designed as a single-arm, two-center, open-label, prospective study. All participants are enrolled in the standard-dose unrelated umbilical cord blood transplantation group to evaluate the efficacy and safety of unrelated umbilical cord blood transplantation in treating Epstein-Barr virus-associated lymphoproliferative disease.

DETAILED DESCRIPTION:
Epstein-Barr virus-associated lymphoproliferative diseases (EBV-LPDs) are a group of disorders characterized by abnormal proliferation of lymphocytes caused by or associated with Epstein-Barr virus (EBV) infection.

Among these, chronic active EBV infection (CAEBV) is a severe systemic EBV-positive lymphoproliferative disease predominantly seen in East Asian populations, especially in Japan, China, and Korea. Unlike in Western countries where B cells are primarily affected, EBV in Asian CAEBV patients mainly infects T cells or NK cells. The clinical manifestations of CAEBV are diverse, including fever, hepatosplenomegaly, lymphadenopathy, rash, and hypersensitivity to mosquito bites. Serious complications include hemophagocytic lymphohistiocytosis (HLH), liver failure, interstitial pneumonia, and coronary artery lesions. Current treatment strategies for CAEBV include immunomodulatory therapy, chemotherapy (including etoposide-containing regimens such as L-DEP, CHOP, etc.), and allogeneic hematopoietic stem cell transplantation. Allogeneic hematopoietic stem cell transplantation (Allo-HSCT) is currently the only potentially curative approach. Patients with severe CAEBV have an extremely poor prognosis without undergoing hematopoietic stem cell transplantation.

EBV-associated lymphomas refer to a category of malignant lymphoid neoplasms driven or implicated in pathogenesis by EBV infection. By infecting B cells, T cells, or NK cells, EBV leads to abnormal cell proliferation and malignant transformation, ultimately resulting in lymphoma. EBV-associated lymphomas are highly heterogeneous, necessitating precise stratification of treatment regimens. For high-risk and refractory EBV-associated lymphomas, allogeneic hematopoietic stem cell transplantation is an effective treatment method.

Allogeneic hematopoietic stem cell transplantation (Allo-HSCT) is a therapeutic procedure that involves the infusion of hematopoietic stem cells from a healthy donor to reconstitute the patient's hematopoietic and immune systems. Numerous international studies have demonstrated that Allo-HSCT is an effective treatment for various EBV-LPDs. Umbilical cord blood transplantation (UCBT) is a specific type of Allo-HSCT. Umbilical cord blood refers to the blood remaining in the umbilical cord and placenta after the cord of a newborn is clamped. This blood is rich in hematopoietic stem cells, and transplantation using this cord blood is termed umbilical cord blood hematopoietic stem cell transplantation.

Given that both the Chinese Expert Consensus on the Diagnosis and Treatment of Chronic Active EBV Disease and international CAEBV management consensuses indicate that Allo-HSCT is currently the only potentially curative method for CAEBV, and considering that internationally published small-sample studies have shown favorable efficacy of UCBT in EBV-LPDs such as CAEBV, data across different disease subtypes remain limited. Therefore, this study aims to further validate the efficacy and safety of unrelated umbilical cord blood transplantation for EBV-associated lymphoproliferative diseases through a single-center, prospective investigation.

ELIGIBILITY:
Inclusion Criteria:General Inclusion Criteria:

All subjects must meet all of the following criteria:

Age range: 14 to 80 years old, inclusive.

Diagnosed with an EBV-associated lymphoproliferative disease (including Chronic Active EBV Infection, EBV-associated Hemophagocytic Lymphohistiocytosis, and EBV-associated Lymphoma).

Meet at least one of the following disease-specific criteria (see below).

ECOG Performance Status score of 0-2 (or Lansky Play-Performance score ≥60 for children).

Expected survival of ≥3 months.

Signed informed consent form (for minors, consent must be provided by a legal guardian).

Disease-Specific Inclusion Criteria:

A. CAEBV Patients: Patients diagnosed with CAEBV according to the 2016 revised WHO classification criteria, who also meet all of the following:

* Persistent or recurrent infectious mononucleosis-like symptoms for more than 3 months.
* Elevated EBV-DNA load in peripheral blood or involved tissues (peripheral blood EBV-DNA > 500 copies/ml).
* Detection of EBV in T or NK cells (via EBER in situ hybridization or LMP1 immunohistochemistry).
* Exclusion of other known immunodeficiency disorders, autoimmune diseases, or neoplastic diseases.

B. EBV-HLH Patients: Meet ≥5 of the HLH-2004 diagnostic criteria:

* Persistent or recurrent infectious mononucleosis-like symptoms for more than 3 months.
* Fever ≥38.5°C.
* Splenomegaly.
* Cytopenias (affecting ≥2 of 3 lineages):
* Hb <90 g/L
* PLT <100 × 10⁹/L
* ANC <1.0 × 10⁹/L
* Hypertriglyceridemia (>3 mmol/L) and/or hypofibrinogenemia (<1.5 g/L).
* Serum ferritin >500 μg/L.
* sCD25 >2400 U/mL.
* Decreased or absent NK cell activity.
* Evidence of hemophagocytosis in bone marrow, spleen, or lymph nodes.

C. EBV-associated Lymphoma Patients:

* Pathologically confirmed diagnosis according to WHO criteria.
* EBV-positive (EBER+).
* Failure of or relapse after first-line therapy.

Exclusion Criteria:Patients meeting any of the following criteria will be excluded:

History of another primary malignancy within 5 years prior to the first treatment.

Uncorrected thyroid dysfunction.

Grade II or higher cardiac disease according to the New York Heart Association (NYHA) classification.

History of organ transplantation.

Planned to receive other types of hematopoietic stem cell transplantation during the study period.

Active infections, including:

Active hepatitis B or hepatitis C.

Positive serum HIV antigen or antibody.

History of syphilis.

Major surgery within 4 weeks prior to the first treatment, or anticipated need for major surgery during the study.

Pregnant or breastfeeding women.

History of severe psychiatric illness or substance abuse.

High risk of complications, such as:

Uncontrolled infection.

Active major visceral hemorrhage.

Known allergy to any component of the investigational drug(s), or a history of severe allergies.

Patients deemed unable to comply with the study procedures and/or follow-up requirements.

-

Ages: 14 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2028-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Overall Response Rate (ORR) | 3 months
  The percentage of patients who achieved complete response (CR) or partial response (PR) after umbilical cord blood transplantation, out of the total number of patients evaluable for efficacy.

SECONDARY OUTCOMES:
Survival | 1 year
  From the date of inclusion to date of death, irrespective of cause Adverse Events
Treatment-Related Adverse Events | through study completion, an average of 1 year
  Adverse events including myelosuppression, liver function damage, infection, bleeding and so on.

CONTACTS AND LOCATIONS:
Overall Officials: Jiexian Ma, Principal Investigator — Huadong Hospital
Locations (2):
- China (2):
  - Huadong hospital, Fudan university, Shanghai, Shanghai Municipality
  - Huashan Hospital, Fudan University, Shanghai, Shanghai Municipality

IPD SHARING:
Plan to Share IPD: Yes
All collected IPD
Supporting Information: Study Protocol, SAP, ICF
Access Criteria: 1 year after completion of this study